CLINICAL TRIAL: NCT04462510
Title: A Comparison Between Ultrasound Guided Ilioinguial/Iliohyphogastic Nerves Block and Infiltration of Wound With Ropivacaine on Post-Operative Pain After Open Repair of Unilateral Inguinal Hernia in Adults: A Randomized Controlled Trial
Brief Title: To Compare Ilioinguinal/Iliohypogastric Block to Wound Infiltration for Pain Relief After Hernia Repair in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Summaiya Ahsan Ali, Principal Investigator, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AgaKhanU1
Record Dates: First submitted 2020-06-07; First posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: To Compare ILI/IHG Block to Wound Infiltration for Pain Relief After Hernia Repair
MeSH Terms: interventions — Dental Occlusion; Anesthesia, Local

STUDY DESIGN:
Intervention Model Description: Single blinded where the patients were blinded. They were randomly divided into local infiltration group or illioinguinal/illiohypograstric block
Who Masked: Participant
Masking Description: The patients were randomized using computer generated numbers and did not know which group did they fall in
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Illioinguinal/Illiohypogastric Block (Experimental): A single shot 20ml of 0.25% Ropivacaine was used to block illioinguinal/illiohypogastric nerves using ultrasound right before incision was given
  Interventions: Procedure: Block/Local infiltration
- Wound infiltration (Experimental): Surgeon infiltrated the wound using 20ml of 0.25% Ropivacaine right after the skin was closed.
  Interventions: Procedure: Block/Local infiltration

INTERVENTIONS:
Procedure: Block/Local infiltration — One group received ILI/IHG Block and the other group received local anesthetic infiltration for pain relief
  Other Names: ILI/IHG Block; Local Infiltration

SUMMARY:
This study was conducted to assess the postoperative painscores in patients undergoing open inguinal hernia repair between two groups receiving either U/S guided ilioinguinal/iliohypogastric nerves block with Ropivacaine or wound infiltration with Ropivacaine.The safety of two analgesic interventions(ilioinguinal/iliohypogastric nerves blocks and wound infiltration) was measured alongwith comparison of opioid use between the two groups over 24 hours postoperatively was made. Patient satisfaction between the two groups was also assessed by the Likert scale.

DETAILED DESCRIPTION:
Pain is a concerning problem in patients with open inguinal hernia repair. Hence, multi modal analgesia is recommended to overcome this issue. Therefore this randomized controlled trial was conducted to compare the analgesic efficacy of ultrasound guided Ilioinguinal/Iliohyphogastric nerve block vs. local anaesthetic infiltration of wound with Ropivacaine on postoperative pain after open repair of unilateral inguinal hernia in adults.

This study was conducted at Aga Khan University Hospital Karachi.It is a Randomised controlled trial conducted from March 2019 to October 2019. 60 participants for elective unilateral open inguinal hernia repair were included. Patients were randomly allocated (30 each) to one of the two groups. Group I received ILI/IHG nerve block where 20mls 0.25% Ropivacaine was infiltrated around the nerves under U/S guidance, and group II received local anaesthetic infiltration (Ropivacaine 20mls 0.25%) at the end of surgery at the incision site to provide postoperative analgesia. Postoperative pain at rest (static) and on movement (dynamic) was assessed on VRS scale at 0= no pain , 1-3=mild pain, 4-6=moderate pain, 7-10=severe pain at 0, 2,6, 12, 24 hours, either in person or telephone. Total tramadol consumption and time for first tramadol requirement was noted.

In addition complications related to IHG block and LA infiltration were observed.Patient satisfaction was also gauged by the LIKERT scale in the questionairre.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between the ages of 18-75 years, scheduled for unilateral open primary hernia repair electively
* American society of Anaesthesiologists(ASA) standard I to IV

Exclusion Criteria:

* BMI below 18 or above 35 kg/m2
* Local anesthetic allergy
* Pregnancy
* Infection at injection site
* Coagulation disorders
* Contraindication to any drug used in the standard anesthesia regimen

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-30 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Pain score | This was measured at 0 hours (immediately) after the surgery
  Pain score was measured using visual analog scale. (VAS). Score of 0-3 was taken as mild pain, 4-6 moderate pain and score of 7-10 was severe pain.
Pain score | This was measured at 2 hours after the surgery
  Pain score was measured using visual analog scale. (VAS). Score of 0-3 was taken as mild pain, 4-6 moderate pain and score of 7-10 was severe pain.
Pain score | This was measured at 6 hours after the surgery
  Pain score was measured using visual analog scale. (VAS). Score of 0-3 was taken as mild pain, 4-6 moderate pain and score of 7-10 was severe pain.
Pain score | This was measured at 12 hours after the surgery
  Pain score was measured using visual analog scale. (VAS). Score of 0-3 was taken as mild pain, 4-6 moderate pain and score of 7-10 was severe pain.
Pain score | This was measured 24 hours after the surgery
  Pain score was measured using visual analog scale. (VAS). Score of 0-3 was taken as mild pain, 4-6 moderate pain and score of 7-10 was severe pain.

SECONDARY OUTCOMES:
Tramadol consumption | This was measured at 0,2,6,12 and 24 hours after the surgery
  Amount of total tramadol consumption was recorded
Patient satisfaction | This was assessed at the end of 24 hours post operatively.
  This was measured on a 5 point Likert scale. A question was asked that 'was the anesthetic care and pain relief effective?' The scale included the options of Strongly disagree, Disagree, Neutral, Agree, Strongly Agree

CONTACTS AND LOCATIONS:
Overall Officials: Summaiya Ali, MBBS, Principal Investigator — Anesthesia Resident
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Khan RI, Hameed M, Ali SA. Comparison of ilioinguial/iliohyphogastic nerves block with woundinfiltration on postoperative pain: A randomised controlled trial. J Pak Med Assoc. 2024 Nov;74(11):1922-1926. doi: 10.47391/JPMA.10859. PMID 39548607